CLINICAL TRIAL: NCT05454020
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dosing, Ascending-Dose Study Evaluating the Safety, Tolerability and Pharmacokinetics of XG004 Applied Topically in Participants With Osteoarthritis of the Knee
Brief Title: A Study of Topical XG004 in Participants With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xgene Pharmaceutical Group (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-XG004-03-OA-01
Record Dates: First submitted 2022-06-16; First posted 2022-07-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (XG004) (Experimental): XG004 in two dose level (5% or 10%) will be applied to the targeted knee
  Interventions: Drug: XG004
- B (Placebo) (Placebo Comparator): Placebo in all cohorts will be applied to the targeted knee.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XG004 — XG004 gel in two concentrations (5% and 10%) will be applied topically once-daily, twice-daily or three times daily in a designated area of the study knee.
  Arms: A (XG004)
Drug: Placebo — Placebo gel will be applied topically once-daily, twice-daily or three times daily in a designated area of the study knee.
  Arms: B (Placebo)

SUMMARY:
This is phase 1 placebo controlled study to evaluate the safety, tolerability and pharmacokinetics of XG004 applied topically in participants with osteoarthritis of the knee

DETAILED DESCRIPTION:
The study will consist of a 4-week Screening period, an 7-day Treatment period and a 7-day Safety follow-up period that will be conducted by telephone for each Cohort.

Up to 32 participants with OA of the knee will be enrolled into 6 cohorts sequentially and assigned treatment on a 3:1 (XG004: placebo) ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 40 to 75 years of age inclusive, at the time of signing the informed consent form.
2. Body Mass Index (BMI) of 18 to 39, inclusive, at the time of Screening visit.
3. Participant who is diagnosed with primary knee OA fulfilling the American College of Rheumatology (ACR) Clinical and Radiographic criteria for ≥ 26 weeks prior to Screening visit.
4. Kellgren-Lawrence Grade II to IV as confirmed by X-ray during Screening visit or within 6 months prior to Screening visit in the study knee.
5. The average daily walking pain scale in the study knee over Day -4 to Day -2 during the Baseline period must be ≥ 4.0 on NRS 0-10 scale.

Exclusion Criteria:

1. Participants with any systemic or dermatological disorder that may interfere with the evaluation of the test site reactions (e.g., atopic dermatitis, contact eczema, psoriasis).
2. Participants with scars, moles, tattoos at application site or other abnormal pigmentation of the skin or skin type that may, in any way, confound interpretation of the study results.
3. Participants with any of the following conditions on the test area: viral (e.g., herpes or varicella) lesions of the skin, fungal or bacterial skin infections, parasitic infections, acne vulgaris, atrophic skin, striae atrophic, fragility of skin veins, ichthyosis, ulcers or wounds.
4. Participants exposed to excessive or chronic ultraviolet (UV) radiation (i.e., sunbathing, solarium); and waxing, laser/IPL hair removal, fake/spray tanning is prohibited 14 days prior to enrollment or who may foresee an intensive UV exposure or swimming during study participation.
5. Known hypersensitivity or allergy to NSAIDs or gabapentinoids or any component(s) of the investigational products. This includes participants exhibiting aspirin or other NSAID-induced symptoms, including bronchospasm, rhinitis, and urticaria or other NSAID-induced allergic symptoms.
6. Participants with unstable or severe illness, including clinically significant malignancy, of hepatic, pulmonary, metabolic, neurologic, cardiovascular, gastrointestinal (e.g., inflammatory bowel disease), hematological, or psychiatric system as indicated on medical history, physical examination, or clinical laboratory, vital signs, and ECG evaluations, or in the opinion of the Investigator.
7. Participants with any report of acute illness or febrile event within 72 hours prior to randomization.
8. Known positive coronavirus disease 2019 (COVID-19) viral test during Screening or within 3 days prior to Day -1, or suspected COVID-19 infection at check-in on Day -1 visit.
9. Participants who cannot refrain from strenuous exercise from 72 hours prior to first study dose through completion of the Safety follow-up visit
10. Any other condition that, in the opinion of the investigator, would jeopardize the safety of the study participant or impact the validity of the study results

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of topical XG004 applied to the study knee in Osteoarthritis (OA) participants through incidence of Treatment Emergent Adverse Events as assessed by CTCAE v5.0 | From baseline to end of treatment up to 14 days

SECONDARY OUTCOMES:
To examine skin response | From day 1 to day 8
  Skin safety and irritability assessment will be conducted after topical application of investigational product. All skin reactions at the applications sites will be examined and scored as per Modified Berger/Bowman Scoring Scale.
  Pain will be examined a 0-10 NRS (numerical rating scale) and higher scores mean a worse outcome.
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments. | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: Maximum concentration (Cmax)
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments. | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: Time to maximum concentration (Tmax)
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: Area under the drug concentration-time curve
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: accumulation ratio (AR)
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: Apparent clearance
To evaluate systemic pharmacokinetic (PK) following topical administration to the knee. Blood will be collected for plasma PK assessments | From baseline to end of treatment up to 8 days
  The following parameter is used for evaluation during PK assessments: Apparent terminal half-life
To explore the penetration of XG004 into the synovial fluid of the knee. Synovial fluid samples will be evaluated for the drug concentrations. | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Guy Ludbrook, Principal Investigator — PARC Clinical research
Locations (1):
- PARC Clinical research, Adelaide, South Australia, Australia